CLINICAL TRIAL: NCT02151474
Title: A Double-Blind, Placebo-Controlled Study Exploring the Safety, Tolerability, and Efficacy of a 28-Day Course of INCB047986 in Subjects With Active Rheumatoid Arthritis
Brief Title: INCB047986 in Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 47986-202
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- INCB047986 4 mg QD (Experimental): INCB047986 4 mg will be orally self-administered once daily (QD) for 28 days.
  Interventions: Drug: INCB047986
- INCB047986 8 mg QD (Experimental): INCB047986 8 mg will be orally self-administered once daily (QD) for 28 days.
  Interventions: Drug: INCB047986
- INCB047986 12 mg QD (Experimental): INCB047986 12 mg will be orally self-administered once daily (QD) for 28 days.
  Interventions: Drug: INCB047986
- INCB047986 placebo QD (Experimental): INCB047986 placebo will be orally self-administered once daily (QD) for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INCB047986
  Arms: INCB047986 12 mg QD; INCB047986 4 mg QD; INCB047986 8 mg QD
Drug: Placebo
  Arms: INCB047986 placebo QD

SUMMARY:
The purpose of this study is to explore the safety, tolerability and efficacy of INCB047986, in subjects with moderate to severe rheumatoid arthritis.

DETAILED DESCRIPTION:
This will be a double-blind, placebo-controlled study with 4 parallel treatment groups. Subjects will be screened for up to 28 days before study drug administration to ensure that all eligibility criteria are met. On Day 1, subjects will be randomized to 1 of 4 dose groups of 15 subjects each (INCB047986 4 mg, 8 mg, 12 mg, or placebo QD). Study drug will be self administered on Days 1 through 28. A follow-up telephone call to the subject to assess safety will occur at Day 42. A final safety and efficacy evaluation will be performed at the Day 58 visit.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 75 years, inclusive.
* Body mass index between 18 and 40 kg/m^2, inclusive.
* Subjects must have a diagnosis of rheumatoid arthritis (RA) of at least 6 months' duration at the time of screening and must satisfy the ACR/European League Against Rheumatism (EULAR) 2010 Classification Criteria (Appendix B).
* Subjects must have active moderate to severe RA as determined by the following:

  * ≥ 6 tender joints (28 joint count),
  * ≥ 4 swollen joints (28 joint count), and
  * CRP level ≥ 6 mg/L.
* Subjects must have a negative tuberculosis (TB) test (QuantiFERON®-TB Gold test or purified protein derivative (PPD)) at screening.

Exclusion Criteria:

* Current or recent history of severe and/or progressive uncontrolled renal, hepatic, hematologic, gastrointestinal, pulmonary, cardiac, neurological, or cerebral disease.
* Current or recent history (< 30 days before screening and/or < 45 days before randomization) of a clinically meaningful bacterial, fungal, parasitic, or mycobacterial infection.
* Onset of RA before the age of 16 years.
* History of known or currently suspected inflammatory disease other than RA
* Current regimen of prednisone or equivalent with an average daily dose of > 10 mg or having been treated with a stable daily dose ≤ 10 mg for < 6 weeks.
* Previous treatment with at Janus kinase (JAK) inhibitor.
* Significant impairment of bone marrow function present at screening
* Receipt of any live vaccine within 2 months before screening or anticipated need for a live vaccine within the 2 months after last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with adverse events, changes in electrocardiograms (ECGs), vital signs, physical examinations, or clinical laboratory evaluations | Baseline through day 28
Percentage of Participants Achieving American College of Rheumatology, 20% Improvement (ACR20) | Baseline through Day 28

SECONDARY OUTCOMES:
Percentage of subjects achieving ACR20 at each visit assessed. | Baseline, Day 8, 15 and Follow-Up
Percentage of subjects achieving American College of Rheumatology, 50% improvement (ACR50) at each visit assessed. | Baseline, Day 8, 15 28 and Follow-Up
Percentage of subjects achieving American College of Rheumatology, 70% improvement (ACR70) at each visit assessed. | Baseline, Day 8, 15 28 and Follow-Up
Change in Disease Activity Score - 28-joint count (DAS28) C-reactive protein (CRP) at the Day 28 visit. | Day 28
Change in DAS28 erythrocyte sedimentation rate (ESR) at the Day 28 visit. | Day 28
Percentage of subjects achieving a DAS28 of ≤ 3.2 at the Day 28 visit. | Day 28
Percentage of subjects achieving a DAS28 of ≤ 2.6 at the Day 28 visit. | Day 28
Change in individual American College of Rheumatology (ACR) assessments. | Day 28
Preliminary pharmacokinetic (PK) | Evaluated after 15 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard Levy, MD, Study Director — Incyte Corporation
Locations (9):
- United States (9):
  - Orange, California
  - DeBary, Florida
  - Palm Harbor, Florida
  - Tampa, Florida
  - Frederick, Maryland
  - Charlotte, North Carolina
  - Oklahoma City, Oklahoma
  - Austin, Texas
  - The Woodlands, Texas